CLINICAL TRIAL: NCT04237064
Title: Photoacoustic Imaging of Atherosclerotic Plaques
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marc van Sambeek (Other)
Collaborators: Eindhoven University of Technology (Other)
Responsible Party: Sponsor-Investigator, Marc van Sambeek, Prof. dr. Marc van Sambeek, Catharina Ziekenhuis Eindhoven
Organization: Catharina Ziekenhuis Eindhoven (Other)
Other Study IDs: R17.029
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Carotid Artery Plaque
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with carotid artery stenosis: In this study, patients in the age of > 18 year will be included that are scheduled for an endarterectomy procedure at CZE.
  Interventions: Diagnostic Test: Photoacoustic imaging

INTERVENTIONS:
Diagnostic Test: Photoacoustic imaging — Photoacoustic imaging

SUMMARY:
Stroke is a major cause of death and disability worldwide. Stenotic carotid arteries can lead to stroke if the cause of the stenosis is a vulnerable atherosclerotic plaque. Recent studies reveal that if a patient has a plaque in the carotid artery it is highly probable that he/she will develop plaques in other superficial arteries like the femoral artery. Currently, duplex ultrasound is used to determine the grade of stenosis and is the main criterion for intervention (endarterectomy) planning. However, the stability, or instability of the plaque cannot be determined non-invasively. Photoacoustics is a novel, non-invasive imaging modality that uses pulsed laser light to generate laser induced ultrasound in the absorbing region of the tissue. Photoacoustic imaging provides optical contrast of biological tissue chromophores with an acoustic resolution and imaging depth, which is promising for visualization of plaque composition. The advantage of photoacoustics is the use of multiple wavelengths, since different tissues respond differently to different wavelengths. Hence, non-invasive, in vivo, morphology assessment is a future application of this new modality that would improve diagnosis and clinical decision making. The drawback is the limited penetration depth of the laser light and the signals generated by surrounding tissue.

A new, integrated photoacoustic device has been developed that meets all safety requirements and has an improved penetration depth, suitable for imaging of carotid arteries with the aim to distinguish between plaques with different morphology.

DETAILED DESCRIPTION:
Objective: The aim of this study is to investigate the feasibility of atherosclerotic plaque imaging using multispectral photoacoustic imaging.

Study design: This is a pilot study where 60 patients with a plaque in one of the carotids, scheduled for an endarterectomy procedure, will be included. Each subject will get a multi-wavelength photoacoustic examination of the carotid plaque. In one group (N = 30), photoacoustic imaging will be performed noninvasively at the TU/e laser lab, which is compliant with laser safety standards, to verify non-invasive, multi-angle, multi-wavelength photoacoustic imaging (Study A). In the second group (N = 30), photoacoustic imaging will be performed pre- and per-operatively (Study B) prior to plaque removal. Here, to ensure a 100% (laser) safe environment, all acquisitions will be performed in the operating theatre. The latter group will be subjected to additional Magnetic Resonance Imaging for validation. After carotid endarterectomie the plaque sample of each patient (Study A and B) will be transported to TU/e for in vitro PA scanning and histology analysis.

Study population: A total of 60 patients with carotid artery disease scheduled for endarterectomy (stenosis grade of > 70% and < 99%).

Intervention (if applicable): endarterectomy (following normal procedure), with an additional photoacoustic image acquisition after incision, before removal of the plaque.

Main study parameters/endpoints: The acoustic (i.e., echographic) and photoacoustic images will be analyzed to determine the ability of distinguishing between different plaque components (intraplaque hemorrhage, lipid pool, vessel wall), examine penetration depth, resolution, and contrast.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must be an adult that is fully competent to give informed consent that has been under surveillance for a plaque in one of the carotid arteries with a stenosis grade between 70 and 99% (based on prior Duplex US examination in the vascular lab) In case of study A, the subject should physically be able to be seated in a chair without moving for 10 to 20 minutes.

Exclusion Criteria:

Minors or incapacitated adults will not be included in the study. Subjects that do not want to participate will also not be included. -

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In this study, patients in the age of > 18 year will be included that are scheduled for an endarterectomy procedure at CZE.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-02-02 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of vulnerable plaque | 2 year
  Demonstration of the feasibility of in vivo photoacoustic imaging of atherosclerotic plaques using multi-angle, multi-wavelength photoacoustics.

CONTACTS AND LOCATIONS:
Overall Officials: Marc RHM van Sambeek, MD PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Hospital Eindhoven, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No